CLINICAL TRIAL: NCT07246629
Title: Prophylactic Use of Intrathecal Calcium Channel Antagonist Through Lumbar Drain in Patients With Subarachnoid Hemorrhage Due to Aneurysmal Rupture
Brief Title: Lumbar Drain With Intrathecal Nicardipine in Aneurysmal Subarachnoid Hemorrhage
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB00139639
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Subarachnoid Hemorrhage
Keywords: cerebral aneurysm; intrathecal nicardipine; vasospasm
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Aneurysm | interventions — Saline Solution; Nicardipine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Sham Comparator): standard treatment of cerebral vasospasm and sham injection of 10 mL preservative-free normal saline in luer-lock sterile syringe
  Interventions: Drug: Normal Saline
- Standard of Care Plus Nicardipine (Experimental): standard treatment of cerebral vasospasm with prophylactic administration of intrathecal nicardipine
  Interventions: Drug: Nicardipine

INTERVENTIONS:
Drug: Normal Saline — 10 mL preservative-free normal saline in luer-lock sterile syringe every 24 hours from randomization through day 14 post-bleed or lumbar drain removal, whichever occurs first.
  Arms: Standard of Care
Drug: Nicardipine — Nicardipine 4 mg will be diluted in preservative-free normal saline to 10 mL in luer-lock sterile syringe every 24 hours from randomization through day 14 post-bleed or lumbar drain removal, whichever occurs first.
  Arms: Standard of Care Plus Nicardipine

SUMMARY:
The purpose of this study is to determine the effectiveness of prophylactic administration of intra-thecal nicardipine though lumbar cerebrospinal fluid drain in prevention of symptomatic vasospasm in patients with subarachnoid hemorrhage due to rupture of cerebral aneurysms.

DETAILED DESCRIPTION:
This is a triple-blinded, prospective, sham, randomized study. The purpose of this research is to determine the effectiveness of prophylactic administration of intra-thecal nicardipine though lumbar cerebrospinal fluid drain in prevention of symptomatic vasospasm in patients with subarachnoid hemorrhage due to rupture of cerebral aneurysms. Patients will be randomized to standard treatment of cerebral vasospasm with prophylactic administration of intrathecal nicardipine vs standard treatment alone. The medication used is FDA approved and will be used through an intra-thecal route through a lumbar drain which is indicated in patients with subarachnoid hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Aneurysmal subarachnoid hemorrhage with Hunt and Hess score 3 or less
* Patient or legal authorized representative available to sign the informed consent form
* Pre-morbid modified Rankin scale of 0 or 1.
* Patients who have lumbar drain placed or planned for cerebrospinal fluid diversion per standard of care
* Patients who are able to be randomized within 72 hours from arrival with aneurysmal subarachnoid hemorrhage or within 24 hours from lumbar drain placement

Exclusion Criteria:

* Pregnant females
* Subarachnoid hemorrhage (SAH) with hunt and hess scale of >3
* SAH due to etiology other than aneurysmal rupture
* Any contraindications in patients receiving calcium channel antagonists like hypersensitivity to dihydropyridines
* Active central nerve infection (CNS) infection or high suspicion of CNS infection
* Hemodynamic instability preventing the use of Nicardipine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Vasospasm | up to hospitalization day 21
  The incidence of symptomatic clinical or radiographic vasospasm in patients treated with prophylactic administration of intrathecal nicardipine though lumbar drain
Incidence of Delayed Cerebral Ischemia | up to hospitalization day 21
  The incidence of symptomatic clinical or radiographic delayed cerebral ischemia in patients treated with prophylactic administration of intrathecal nicardipine though lumbar drain

SECONDARY OUTCOMES:
Modified Rankin Scale Score | month 6
  The Modified Rankin Scale is a clinical tool used to assess the functional disability after a stroke. It is a six-point ordinal scale that measures the patient's ability to perform activities of daily living. Score Range: 0 no symptoms, 1 no significant disability, 2 slight disability, 3 moderate disability, 4 moderately severe disability, 5 severe disability, 6 dead.
Incidence of Meningitis | up to hospitalization day 21
  Incidence of meningitis as confirmed by clinical and laboratory findings

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Joshi, MD, Principal Investigator — Advocate Lutheran General Hospital
Locations (1):
- Advocate Lutheran General Hospital, Park Ridge, Illinois, United States

IPD SHARING:
Plan to Share IPD: No